CLINICAL TRIAL: NCT05062200
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-77242113 in Healthy Japanese Participants and a Single Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-77242113 in Healthy Chinese Participants
Brief Title: A Study of JNJ-77242113 in Healthy Japanese and Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR109097; 77242113PSO1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: JNJ-77242113 or Placebo (Single Ascending Dose [SAD]) (Experimental): Japanese participants will receive single oral dose 1 of JNJ-77242113 (immediate-release [IR] tablet) or matching placebo on Day 1 in Cohort 1 of Part 1.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Cohort 2: JNJ-77242113 or Placebo (SAD) (Experimental): Japanese participants will receive single oral dose 2 of JNJ-77242113 (IR tablet) or matching placebo on Day 1 in Cohort 2 of Part 1.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Cohort 3: JNJ-77242113 or Placebo (Single Dose [SD]) (Experimental): Chinese participants will receive single oral dose 2 of JNJ-77242113 (IR tablet) or matching placebo on Day 1 in Cohort 3 of Part 2.
  Interventions: Drug: JNJ-77242113; Drug: Placebo
- Cohort 4: JNJ-77242113 or Placebo (SD) (Experimental): Japanese participants will receive single oral dose 3 of JNJ-77242113 (delayed-release [DR] tablet) with absorption enhancer (AbE) or matching placebo on Day 1 in Cohort 4 of Part 3.
  Interventions: Drug: JNJ-77242113; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 will be administered as an oral tablet.
Drug: Placebo — Matching placebo will be administered as an oral tablet.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of JNJ-77242113 after single ascending oral dose administration as an immediate-release (IR) tablet formulation in healthy Japanese participants and after single oral dose administration as an IR tablet formulation in healthy Chinese participants; and as a delayed release (DR) tablet formulation in healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* For Parts 1 and 3: Japanese male or female of non-childbearing potential, who have parents and maternal and paternal grandparents who are of Japanese ethnicity
* For Part 2: Chinese male or female of non-childbearing potential, who have parents and maternal and paternal grandparents who are of Chinese ethnicity
* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the study population. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body weight not less than 50 kilograms (kg) and body mass index within the range 18 and 30 kilograms per meter square (kg/m^2) (inclusive)
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted

Exclusion Criteria:

* History of malignancy before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Known allergies, hypersensitivity, or intolerance to JNJ-77242113 or its excipients
* Use of a live vaccine within 30 days prior to screening or anticipated need for a live vaccine during the study or for 30 days following the dose of study drug
* Received an experimental drug (including investigational vaccines) or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the dose of the study intervention is scheduled
* Test positive for human immunodeficiency virus (HIV)-1 and 2 antigen/antibodies, test positive for hepatitis C antibodies, test positive for syphilis, or test positive for hepatitis B virus (HBV) infection at screening

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Parts 1, 2 and 3: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 6 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Parts 1, 2 and 3: Plasma Concentration of JNJ-77242113 | Predose up to 48 hours postdose (Up to Day 3)
  Plasma samples will be analyzed to determine concentrations of JNJ-77242113 using a validated, specific and sensitive method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency